CLINICAL TRIAL: NCT03411252
Title: Mirabegron in Achalasia: A Clinical and Manometric Proof of Concept Pilot Study
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: inability to enroll
Sponsor: Thomas Jefferson University (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, Jeff GI, Dr Anthony J DiMarino, Chair, Division of Gastroenterology, Thomas Jefferson University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17P.054
Record Dates: First submitted 2017-12-11; First posted 2018-01-26 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Achalasia
MeSH Terms: conditions — Esophageal Achalasia | interventions — mirabegron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Mirabegron (Experimental): Patients will receive 50 mg of oral Mirabegron daily for 4 weeks and then switch to placebo by mouth daily for an additional 4 weeks.
  Interventions: Drug: Mirabegron 50 MG; Drug: Placebo
- Placebo (Placebo Comparator): Patients will receive placebo by mouth daily for 4 weeks and then switch to oral Mirabegron 50 mg daily for an additional 4 weeks.
  Interventions: Drug: Mirabegron 50 MG; Drug: Placebo

INTERVENTIONS:
Drug: Mirabegron 50 MG — Myrbetriq (Mirabegron) tablet
  Other Names: Myrbetriq
Drug: Placebo — Sugar pill manufactured to mimic Mirabegron
  Other Names: Placebo (for Mirabegron)

SUMMARY:
This study evaluates whether a medication called mirabegron is better than placebo (sugar pill) in helping patients with achalasia swallow better. Each patient will receive either mirabegron or the placebo for 4 weeks followed by the opposite medication. Each patient will complete several surveys and undergo several tests to determine if the mirabegron is helping reduce the pressures in the esophagus (swallowing tube).

DETAILED DESCRIPTION:
Achalasia is characterized by incomplete or absent relaxation of the lower esophageal sphincter (LES) and loss of esophageal peristalsis which leads to dysphagia. Standard of care for achalasia includes endoscopic management (dilation and injection of injection of botulinum toxin) and surgery, however both of these options carry procedural risks, may lose efficacy over time and many patients are not appropriate candidates for these treatment options. Unfortunately, there are limited oral medications for patients with achalasia. Mirabegron is an oral beta-3 agonist currently FDA approved for overactive bladder that works by relaxing the bladder muscles. Beta-3 receptors have also been identified in the LES with stimulation leading to LES relaxation in preclinical studies. Through a proof of concept pilot study, the investigators aim to evaluate the effect of mirabegron in patients with achalasia via high resolution manometry and a validated dysphagia scale.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old < Age < 75 years old with prior diagnosis of achalasia via manometry and/or radiographically

Exclusion Criteria:

* < 18 years old or > 75 years old
* History of hypertension not controlled on oral medications (blood pressure > 160/100 mm Hg)
* No prior history of hypertension with a blood pressure > 160/100 mm Hg
* History of bladder outlet obstruction
* History of angioedema
* Pregnant or breast-feeding women: Women between 18 and 40 years old who are enrolled in the study will be required to use a form of birth control during the study
* Patients currently receiving certain medications (digoxin, warfarin, any overactive bladder medications, thioridazine, flecainide, propafenone, phosphodiesterase inhibitors)
* Patients with prolonged QTc interval or risk factors to develop it:

  * Baseline QTc on EKG of > 450 milliseconds
  * History of additional risk factors for Torsades de Pointes (heart failure, family history of long QT syndrome)
  * Concomitant medications that prolong the QTc interval: ranolazine, sotalol, dofetilide, procainamide, disopyramide, propafenone, azole antifungals, fluoroquinolones, macrolide antibiotics, HIV antiretrovirals, chemotherapy, beta-2 agonists, tricyclic antidepressants, selective serotonin reuptake inhibitors
* Prior surgeries for achalasia
* < 2 months since last endoscopic botulinum toxin injection into LES or endoscopic dilation
* Stage 4 Chronic kidney disease (severe renal impairment with GFR 15-29 ml/min), Stage 5 Chronic Kidney disease (GFR < 15 ml/min or on dialysis)
* Childs Pugh B (moderate) or C (severe) Cirrhotic (hepatic impairment)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Changes in lower esophageal sphincter pressures | Change in lower esophageal sphincter pressure from baseline after 4 weeks of placebo or Mirabegron
  Evaluation of changes in lower esophageal sphincter pressures using high resolution manometry

SECONDARY OUTCOMES:
Eckardt Achalasia Score (EAS) | Patients will complete the EAS on study day -14, 0, 7, 28, 42, 49, 70, 84. We will evaluate changes in patient's EAS between day 0 and all of these time points.
  Patients will complete the Eckardt Achalasia score which is a simple written scale evaluating dysphagia, regurgitation, retrosternal pain and weight loss. Patients report their symptoms from a 0 to 3. Weight loss (0-none, 1: < 5 kg, 2: 5-10 kg, 3: > 10 kg), Dysphagia (0-none, 1-occasional, 2-daily, 3-each meal), Retrosternal pain (0-none, 1-occasional, 2-daily, 3-each meal), Regurgitation (0-none, 1-occasional, 2-daily, 3-each meal). The value for each of the 4 categories is added together to give the EAS. This EAS will be reported for each time point below. A higher score is consistent with worse achalasia and worse outcomes. A lower score is consistent with less severe achalasia and better outcomes. The total range is 0 (no symptoms) to 12 (severe symptoms). There are no subscales.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No